CLINICAL TRIAL: NCT05546411
Title: A Phase 2 Study of Neoadjuvant NIS793 in Combination With mFOLFIRINOX in Resectable and Borderline Resectable Pancreatic Adenocarcinoma (PDAC)
Brief Title: A Trial of NIS793 With FOLFIRINOX in Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Novartis, the drug manufacturer of NIS793, notified Dana Farber Cancer Institute that they are stopping all clinical development of NIS793 in pancreatic cancer, effective immediately.
Sponsor: Kimberly Perez, MD (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Kimberly Perez, MD, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-314
Record Dates: First submitted 2022-09-07; First posted 2022-09-19 (Actual); Results first posted 2024-07-16 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-11

CONDITIONS: Pancreatic Cancer; Resectable Pancreatic Cancer; Borderline Resectable Pancreatic Adenocarcinoma; Pancreatic Adenocarcinoma
Keywords: Pancreatic Cancer; Resectable Pancreatic Cancer; Borderline Resectable Pancreatic Adenocarcinoma; Pancreatic Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Fluorouracil; Oxaliplatin; Irinotecan; Leucovorin; NIS-793; Chemoradiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- mFOLFIRINOX + NIS793 (Experimental): Participants will be randomly assigned to receive:
  * FOLFIRINOX + NIS793 on day 1 of each 14 day cycle up to 8 cycles/16 weeks
  * Cycles 9+: Based on study team determination, some participants may be offered chemoradiation following completion of chemotherapy and/or surgery following either completion of chemotherapy or chemoradiation
  Interventions: Drug: mFOLFIRINOX; Drug: 5-Fluorouracil (5-FU); Drug: Oxaliplatin; Drug: Irinotecan; Drug: Leucovorin; Drug: NIS793; Radiation: Chemoradiation; Procedure: Surgery
- mFOLFIRINOX (Active Comparator): Participants will be randomly assigned to receive:
  * FOLFIRINOX on day 1 of each 14 day cycle up to 8 cycles/16 weeks
  * Cycles 9+: Based on study team determination, some participants may be offered chemoradiation following completion of chemotherapy and/or surgery following either completion of chemotherapy or chemoradiation
  Interventions: Drug: mFOLFIRINOX; Drug: 5-Fluorouracil (5-FU); Drug: Oxaliplatin; Drug: Irinotecan; Drug: Leucovorin; Radiation: Chemoradiation; Procedure: Surgery

INTERVENTIONS:
Drug: mFOLFIRINOX — Combination of the drugs 5-Fluorouracil (5-FU), Oxaliplatin, Irinotecan, and Leucovorin given by intravenous infusion
Drug: 5-Fluorouracil (5-FU) — Part of the FOLFIRINOX drug combination, given by intravenous infusion
  Other Names: Adrucil
Drug: Oxaliplatin — Part of the FOLFIRINOX drug combination, given by intravenous infusion
  Other Names: Eloxatin
Drug: Irinotecan — Part of the FOLFIRINOX drug combination, given by intravenous infusion
  Other Names: Camptosar; Camptothecin-11; CPT-1
Drug: Leucovorin — Part of the FOLFIRINOX drug combination, given by intravenous infusion
  Other Names: Calcium Leucovorin; Citrovorum Factor; Folinic Acid
Drug: NIS793 — Given by intravenous infusion
  Arms: mFOLFIRINOX + NIS793
Radiation: Chemoradiation — Combination of Chemo (Capecitabine) and Radiation Therapy
Procedure: Surgery — Surgical removal of tumor

SUMMARY:
This study is being done to evaluate the safety and efficacy of adding NIS793 to standard of care FOLFIRINOX treatment for pancreatic cancer.

The names of the study interventions involved in this study are:

* NIS793
* FOLFIRINOX (Folinic acid/Leucovorin, 5-Fluorouracil, Irinotecan, and Oxaliplatin)

Other interventions may include:

* Chemoradiation Therapy
* Surgery

DETAILED DESCRIPTION:
This is a randomized phase 2 study evaluating the efficacy of NIS793, a TGF-beta inhibitor, when added to a standard chemotherapy program of modified FOLFIRINOX for people with previously-untreated, resectable or borderline resectable pancreatic adenocarcinoma.

The U.S. Food and Drug Administration (FDA) has not approved NIS793 as a treatment for any disease. NIS793 works by blocking a molecule called TGF-beta. TGFbeta has been shown to promote the growth of pancreatic cancer and this study is examining if the addition of a TGF-beta blocking drug will allow the chemotherapy to work better against the cancer.

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

Participants will be randomized into two groups of:

* Arm A will receive standard chemotherapy, mFOLFIRINOX, in combination with NIS793.
* Arm B will receive standard chemotherapy, mFOLFIRINOX.

Based on study team determination, some participants may be offered chemoradiation following completion of chemotherapy and/or surgery following either completion of chemotherapy or chemoradiation.

Study treatment is expected to last up to 16 weeks unless disease symptom worsens .

It is expected that about 45 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* The clinical, radiographic, and pathologic evidence support a diagnosis of pancreatic adenocarcinoma, with histology confirmatory for adenocarcinoma.
* Subjects must be determined to meet the criteria for resectable or borderline resectable pancreatic cancer based on the M.D. Anderson Cancer Center (MDACC) and Alliance Intergroup Criteria classification at initial diagnosis (Table 1). Patients with locally advanced or metastatic disease are not eligible for this trial.
* Criteria for resectability of pancreatic cancer

  * Vessel: SMA, Resectable: No extension; normal fat plane between the tumor and the artery, Borderline resectable: Interface between tumor and vessel measuring less than 180º of the circumference of the vessel wall, Locally advanced (Not Eligible): Encased (>180°)
  * Vessel: Celiac axis, Resectable: No extension, Borderline resectable: Interface between tumor and vessel measuring less than 180º of the circumference of the vessel wall, Locally advanced (Not Eligible): Encased and no technical option for reconstruction usually because of extension to the celiac axis/ splenic/left gastric junction or the celiac origin
  * Vessel: Common hepatic artery, Resectable: No extension, Borderline resectable: Reconstructable§, short-segment interface between tumor and vessel of any degree, Locally advanced (Not Eligible): Encased and no technical option for reconstruction usually because of extension to the celiac axis/ splenic/left gastric junction or the celiac origin Vessel: SMV/PV, Resectable: Patent, Borderline resectable:SMV/PV Patent Interface between tumor and vessel measuring 180º or greater of the circumference of the vessel wall, and/or reconstructable§ occlusion Occluded and no technical option for reconstruction, Locally advanced (Not Eligible): Occluded and no technical option for reconstruction

    * Referenced from: Varadhachary et al., 2006(6) and Katz et al, 2013 (8). SMA, superior mesenteric artery; SMV/PV, superior mesenteric vein/portal vein.
    * Normal vein or artery proximal and distal to the site of suggested tumor-vessel involvement suitable for vascular reconstruction
* In subjects requiring biliary decompression, biliary stent or drainage using percutaneous transhepatic cholangiogram (PTC) are allowed.
* Participants must be ≥18 years of age at the time of enrollment.
* Participants must have an ECOG performance status 0-1 (see Appendix A).
* Participants must have adequate organ and marrow function as defined as:

  * Absolute neutrophil count ≥1,500/mcL
  * Platelets ≥100,000/mcL
  * Total bilirubin ≤1.5 × institutional upper limit of normal
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
  * Creatinine ≤1.5 × institutional upper limit of normal OR
  * Creatinine clearance ≥60 mL/min/1.73 m2 for participants with creatinine levels above 1.5 × upper limit of normal. Creatinine clearance can be calculated per institutional standard.
* Female subjects of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity for the course of the study through 9 months after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study therapy.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Has locally advanced or metastatic disease as determined by CT scan or MRI.
* Tumors with histologic features in addition to an adenocarcinoma component are excluded. Variant histologies include but are not limited to adenosquamous, squamous, neuroendocrine, undifferentiated with osteoclast like giant cells, acinar, hepatoid, medullary carcinomas.
* Has either had any prior chemotherapy or targeted small molecule therapy, or immunotherapy or radiation therapy for pancreatic cancer.

Note: If subject received major surgery for reason other than pancreatic cancer they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.

* Has a known prior or current synchronous malignancy, except:

  * Malignancy that was treated with curative intent and for which there has been no known active disease for >5 years prior to enrollment
  * Curatively treated non-melanoma skin cancer, cervical cancer in situ or prostatic intraepithelial neoplasia, without evidence of prostate cancer.
* Significant history of uncontrolled cardiac disease defined as uncontrolled hypertension (defined by a systolic BP >=160 mm Hg and/or diastolic BP >= 100mm Hg), unstable angina, myocardial infarction within the last 4 months, or uncontrolled congestive heart failure. Subjects with a history of cardiac disease should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants should be class 2B or better.
* Has a medical history or current diagnosis of myocarditis.
* Has a left ventricular ejection fraction <50%, cardiac valvulopathy > grade 2, or elevated cardiac enzymes (troponin I) elevation > 2x ULN.
* Has a condition/s that are considered to have a high risk of clinically significant GI bleed or any other condition associated with or history of significant bleeding.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Patients receiving physiological replacement doses of corticosteroids (10mg of prednisone or equivalent) are allowed.
* Has known active, uncontrolled HIV (high viral load), Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).

  * Patients who have been vaccinated for hepatitis B and do not have a history of infection are eligible.
* Has received a live vaccine within 30 days prior to the first dose of trial treatment. COVID-19 vaccination or booster is permitted any time prior to enrollment or during treatment on trial, in a manner consistent with individual institutional guidelines.
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.
* Has an active serious infection requiring systemic therapy.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Subject is unable or unwilling to participate in a study related procedure.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-01-06 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Perez, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- mFOLFIRINOX + NIS793: Participants will be randomly assigned to receive:
  * FOLFIRINOX + NIS793 on day 1 of each 14 day cycle up to 8 cycles/16 weeks
  * Cycles 9+: Based on study team determination, some participants may be offered chemoradiation following completion of chemotherapy and/or surgery following either completion of chemotherapy or chemoradiation
  mFOLFIRINOX: Combination of the drugs 5-Fluorouracil (5-FU), Oxaliplatin, Irinotecan, and Leucovorin given by intravenous infusion
  5-Fluorouracil (5-FU): Part of the FOLFIRINOX drug combination, given by intravenous infusion
  Oxaliplatin: Part of the FOLFIRINOX drug combination, given by intravenous infusion
  Irinotecan: Part of the FOLFIRINOX drug combination, given by intravenous infusion
  Leucovorin: Part of the FOLFIRINOX drug combination, given by intravenous infusion
  NIS793: Given by intravenous infusion
  Chemoradiation: Combination of Chemo (Capecitabine) and Radiation Therapy
  Surgery: Surgical removal of tumor
- mFOLFIRINOX: Participants will be randomly assigned to receive:
  * FOLFIRINOX on day 1 of each 14 day cycle up to 8 cycles/16 weeks
  * Cycles 9+: Based on study team determination, some participants may be offered chemoradiation following completion of chemotherapy and/or surgery following either completion of chemotherapy or chemoradiation
  mFOLFIRINOX: Combination of the drugs 5-Fluorouracil (5-FU), Oxaliplatin, Irinotecan, and Leucovorin given by intravenous infusion
  5-Fluorouracil (5-FU): Part of the FOLFIRINOX drug combination, given by intravenous infusion
  Oxaliplatin: Part of the FOLFIRINOX drug combination, given by intravenous infusion
  Irinotecan: Part of the FOLFIRINOX drug combination, given by intravenous infusion
  Leucovorin: Part of the FOLFIRINOX drug combination, given by intravenous infusion
  Chemoradiation: Combination of Chemo (Capecitabine) and Radiation Therapy
  Surgery: Surgical removal of tumor
Period: Overall Study
Arm/Group | mFOLFIRINOX + NIS793 | mFOLFIRINOX
Started | 6 | 2
Completed | 4 | 1
Not Completed | 2 | 1
Not completed — Progressive Disease | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Metastatic disease | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | mFOLFIRINOX + NIS793 | mFOLFIRINOX | Total
Number analyzed (Participants) | 6 | 2 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 1 | 5
  >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 5 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 2 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 2 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Major Pathological Response Rate (MPR)
Description: Major pathological response (MPR) defined as <5% residual tumor cells visible in the pancreatic resection specimen. The major pathological response rate will be analyzed among all patients who start protocol therapy, including those not resected due to early progression, death or off study.
Time Frame: Pathology review is done in surgery assessments, once within 14 days prior to the operation.
Population: This study was closed prematurely by the drug manufacturer, Novartis, due to safety concerns. At the time of study closure, 8 patients had received any protocol therapy. Out of the 8 participants who received treatment, only 5 underwent surgery before study closure.
Measure: Count of Participants; unit: Participants
Arm/Group | mFOLFIRINOX + NIS793 | mFOLFIRINOX
Number analyzed (Participants) | 6 | 2
Participants | 0 | 0

2. Secondary Outcome: Treatment-Related Toxicity Rate
Description: All adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv5 as reported on case report forms will be counted. Rate is the proportion of treated participants experiencing at least one treatment-related AE of any type during the time of observation.
Time Frame: Cycle 1 Day 1 through 30 days post last treatment date, up to 9 months.
Population: This study was closed prematurely by the drug manufacturer, Novartis, due to safety concerns. At the time of study closure, 6 patients had received mFOLFIRINIX + NIS793 (Arm A) protocol therapy and 2 received mFOLFIRINOX (Arm B).
Measure: Count of Participants; unit: Participants
Arm/Group | mFOLFIRINOX + NIS793 | mFOLFIRINOX
Number analyzed (Participants) | 6 | 2
Participants | 5 | 0

3. Secondary Outcome: Median Progression-free Survival (PFS)
Description: Progression-free survival based on the Kaplan-Meier method is defined as the duration of time from study entry to documented disease progression (PD) or death. Per RECIST 1.1 criteria: progressive disease (PD) is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions.
Time Frame: From randomization (or registration) to the earlier of progression or death due to any cause, up to 9 months. Participants alive without disease progression are censored at date of last disease evaluation.
Population: 4 participants received scans for PFS analysis in Arm A and 1 participant received a scan for PFS analysis in Arm B.
Measure: Median (Full Range); unit: days
Arm/Group | mFOLFIRINOX + NIS793 | mFOLFIRINOX
Number analyzed (Participants) | 4 | 1
days | 114 [108 to 118] | 122 [122 to 122]

4. Secondary Outcome: Median Overall Survival (OS)
Description: OS is based on the Kaplan-Meier method, defined as the time from study entry to death or censored at date last known alive.
Time Frame: Post treatment follow up done at least once every 12 weeks (+/- 28 days), up to 9 months.
Population: All participants were analyzed from the date of study entry until the date the participant came off study. No deaths were recorded while the participants were on study. All dates reflect the date the study was terminated or the date a subject began a new therapy and therefore transitioned off study.
Measure: Median (Full Range); unit: days
Arm/Group | mFOLFIRINOX + NIS793 | mFOLFIRINOX
Number analyzed (Participants) | 6 | 2
days | 184 [43 to 254] | 155.5 [85 to 226]

ADVERSE EVENTS:
Time Frame: Adverse events were reviewed and reported after the initial dose of study treatment, during treatment, or within 30 days of the last dose of treatment. Adverse events were recorded between the first patient treated (February 2023) and 30 days out from the last patient ending treatment (October 2023), equaling a collection time of 9 months.
Arm/Group | mFOLFIRINOX + NIS793 | mFOLFIRINOX
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/6 | 2/2
Other Adverse Events (participants affected / at risk) | 6/6 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | mFOLFIRINOX + NIS793 (N=6) | mFOLFIRINOX (N=2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | mFOLFIRINOX + NIS793 (N=6) | mFOLFIRINOX (N=2)
Anemia (Blood and lymphatic system disorders) | 5 (8) | 1 (8)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (5)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (5) | 2 (5)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (2)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 4 (8) | 1 (4)
Thrush (Infections and infestations) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (3) | 1 (1)
Alkaline phosphatase increased (Investigations) | 4 (6) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Cardiac troponin I increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 2 (3) | 2 (4)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 4 (4) | 0 (0)
Paresthesia (Nervous system disorders) | 4 (5) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nail changes (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-13): https://cdn.clinicaltrials.gov/large-docs/11/NCT05546411/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-02): https://cdn.clinicaltrials.gov/large-docs/11/NCT05546411/ICF_001.pdf